CLINICAL TRIAL: NCT06855329
Title: PRIME-PPF: PRospective phenotypIng and Multi-omic Endotyping of Progressive Pulmonary Fibrosis
Brief Title: PRospective phenotypIng and Multi-omic Endotyping of Progressive Pulmonary Fibrosis
Acronym: PRIME-PPF
Status: Recruiting | Type: Observational
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: University of Michigan (Other); University of Virginia (Other); Johannes Gutenberg University Mainz (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Fernando J Martinez, Professor, University of Massachusetts, Worcester
Other Study IDs: STUDY00002006
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Progressive Pulmonary Fibrosis; Interstitial Lung Disease
Keywords: Progressive pulmonary fibrosis; Interstitial lung disease; PRIME; PRIME-PPF; PPF
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, serum, DNA, RNA, nasal, buccal, and fecal swabs
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective, observational cohort study. Participants with non-idiopatic pulmonary fibrosis, interstitial lung disease (ILD) will be followed for 24 months to systematically collect clinical, imaging, and biospecimen data. The primary objective is to optimize progressive pulmonary fibrosis (PPF) classification and establish PPF incidence for key ILD subtypes. Additional exploratory objectives are to 1) Prospectively validate a novel PPF classifier and assess performance durability over time, and 2) Determine whether multi-dimensional PPF prediction outperforms component approaches.

DETAILED DESCRIPTION:
This is a prospective, cohort study with no study investigational therapy prescribed. Patients with non-idiopathic pulmonary fibrosis (non-IPF) fibrosing ILD, including connective tissue disease associated ILD (CTD-ILD), fibrotic hypersensitivity pneumonitis (fHP) and non-IPF idiopathic interstitial pneumonia (IIP) will be recruited. Consented participants with non-IPF ILD will be carefully phenotyped with extensive clinical, physiological, and imaging data. After confirmation of eligibility, participants will undergo protocolized follow-up over 24 months. Clinical data and blood biospecimens will be collected at protocolized time points throughout the study.

The primary outcome is 12-month transplant-free survival (TFS), following a 12-month observation period with TFS defined as the time from 12-month PFT to death, lung transplant or censoring at 12 months or earlier if lost to follow-up. This research will determine whether a ≥10% relative decline in FVC occurring during the 12-month observation period is associated with TFS over the subsequent 12 months. The investigators will then explore other proposed PPF criteria using the same approach. Additionally, the investigators will determine test performance characteristics of a novel proteomic biomarker for predicting PPF at 12 months and compare performance of this classifier to a multi-dimensional approach that incorporates clinical data and quantitative CT data.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years with a diagnosis of non-IPF fibrosing ILD due to CTD-ILD, fHP, or non-IPF IIP based on central review
* Diagnosis of Fibrotic ILD as determined by site investigator.
* Willingness to comply with study procedures and follow-up.
* Provide written informed consent.

Exclusion Criteria:

* Site diagnosis of fibrosing ILD >5 years prior to Visit 1 (Screening and Baseline Visit).
* Minimal ILD, defined as reticular opacities and/or ground-glass opacities without architectural distortion (traction bronchiolectasis/bronchiectasis or honeycombing) affecting < 5% of the lung on centralized evaluation of HRCT at Visit 1 (Screening and Baseline Visit). High quality historical chest HRCT may be used if performed within 90 days prior to Visit 1.
* Extent of emphysema >15% of total lung volume or greater than extent of fibrosis based on central, qualitative assessment of HRCT at Visit 1. High quality historical chest HRCT may be used if performed within 90 days prior to Visit 1.
* Active malignancy within one year prior to Visit 1 (except for non-melanoma skin cancer requiring local treatment).
* Inability to complete full PFT (spirometry and DLCO) at Visit 1. Historical PFT may be used if performed within 90 days prior to Visit 1.
* Taking nintedanib or nerandomilast at Visit 1.
* Pregnancy at screening or plans to become pregnant during follow-up.
* Participation in an interventional clinical trial for fibrotic ILD at the time of Visit 1, or receipt of an investigational drug within the previous 4 weeks of the enrollment visit (Visit 1) or 5 times the half-life, if longer.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with non-idiopathic pulmonary fibrosis (non-IPF) fibrosing ILD, including connective tissue disease associated ILD (CTD-ILD), fibrotic hypersensitivity pneumonitis (fHP) and non-IPF idiopathic interstitial pneumonia (IIP).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Transplant-free survival (TFS) | 12-months to 24-months (following an observation period from 0 months to 12 months)
  TFS is defined as the time from the 12-month pulmonary function tests to death or lung transplant.
  Censoring will occur at 12-months or earlier if lost to follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Martinez, MD, MS, Principal Investigator — University of Massachusetts Chan Medical School; Justin Oldham, MD, MS, Principal Investigator — University of Michigan; Cathie Spino, DSc, Principal Investigator — University of Michigan; Imre Noth, MD, MS, Principal Investigator — University of Virginia; Michael Kreuter, MD, Principal Investigator — Johannes Gutenberg University Mainz; Dinesh Khanna, MD, MS, Principal Investigator — University of Michigan; Luca Richeldi, MD, PhD, Principal Investigator — Policlinico Gemelli
Locations (13):
- United States (5):
  - University of Massachusetts Chan Medical School, Worcester, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - University of Texas Southwestern, Dallas, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Prince Charles Hospital, Brisbane, Queensland
  - Austin Health, Melbourne, Victoria
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of British Columbia, Vancouver, British Columbia
- University College Dublin, Dublin, Ireland, Ireland
- United Kingdom (2):
  - Royal Brompton, London, Greater London
  - University Hospital Southampton, Southampton, Hampshire

IPD SHARING:
Plan to Share IPD: No